CLINICAL TRIAL: NCT06294197
Title: Examination of the Effects of Pelvic Floor Exercises on Vaginal and Sexual Health in Postmenopausal Women.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hatice Gulsah Kurne (Other)
Responsible Party: Sponsor-Investigator, Hatice Gulsah Kurne, Student, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PhD Thesis
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Sexual Dysfunction; Postmenopausal Symptoms; Pelvic Floor Muscle Weakness
Keywords: Postmenopause; vagina; vaginal dryness; sexual function; dyspareunia; quality of life
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Dyspareunia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized Healthy Participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Exercises (Experimental): In the intervention types, women are given training on pelvic floor exercises, that they can perform in the form of home exercises for 12 weeks. Before starting pelvic floor exercises therapy, a physiotherapist who specializes in pelvic floor compatibility will provide information about the location of the pelvic floor muscles through anatomical models and their effect on healthy, vaginal and sexual function. The effects of pelvic floor exercises on this system will be explained on an individual basis, and normal palpation is required to demonstrate their correct execution of contraction of the pelvic floor muscles. Participants will be taught how to contract and contract different muscles, such as the abdominal muscles, hip muscles, and gluteal muscles, or how to avoid pelvic tilt during contraction, and how to perform both rapid and sustained contractions.
  Interventions: Other: Pelvic Floor Exercises
- Control (No Intervention): No intervention will be made in the control unit.

INTERVENTIONS:
Other: Pelvic Floor Exercises — In the intervention types, women are given training on pelvic floor exercises, that they can perform in the form of home exercises for 12 weeks. Before starting pelvic floor exercises therapy, a physiotherapist who specializes in pelvic floor compatibility will provide information about the location of the pelvic floor muscles through anatomical models and their effect on healthy, vaginal and sexual function. The effects of pelvic floor exercises on this system will be explained on an individual basis, and normal palpation is required to demonstrate their correct execution of contraction of the pelvic floor muscles. Participants will be taught how to contract and contract different muscles, such as the abdominal muscles, hip muscles, and gluteal muscles, or how to avoid pelvic tilt during contraction, and how to perform both rapid and sustained contractions.
  Other Names: Pelvic Floor Muscle Training
  Arms: Pelvic Floor Exercises

SUMMARY:
The purpose of this study; To investigate the effects of pelvic floor muscle exercises on vaginal and sexual health in postmenopausal women. Vaginal symptoms such as vaginal dryness, burning and dyspareunia occur in the postmenopausal period. Vaginal symptoms affect sexual function, leading to a decrease in quality of life. In our study, we plan to evaluate vaginal dryness, one of the vaginal symptoms, using Schirmer's Test. Also in our study; Severities of vaginal dryness, burning and dyspareunia will be evaluated with the visual analog scale (VAS), sexual function will be evaluated with the Post-Menopausal Sexuality Questionnaire and Female Sexual Function Scale, vaginal aging will be evaluated with the Daily Effect of Vaginal Aging Scale, and the presence/severity of pelvic floor symptoms will be evaluated with the Pelvic Floor Distress Inventory-20. The cases will be randomized into two groups and pelvic floor exercises will be given to one group. After the exercises are given, vaginal pH and moistness will be evaluated for acute effect. In the other group, vaginal PH and moisture will be measured after 5 minutes. The cases will be followed without any intervention to the control group. After 12 weeks, the same evaluations will be made to both groups and the results will be compared. The data will be compared using appropriate statistical methods (statistical significance value will be taken as p<0.05) and discussed with the literature.

DETAILED DESCRIPTION:
The World Health Organization defines menopause as the permanent cessation of menstruation due to excessive loss of follicular parts (1). "Menopause" terminologically refers to the last menstrual cycle. The "postmenopause" period follows the last menstrual cycle and continues to restrict the 12-month period of amenorrhea (2). During the menopausal period, signs and symptoms of formation may occur in structures sensitive to care (labia major/minor, clitoris, introitus, vagina, urethra and environments). These signs and symptoms include normal dryness, irritation of the vulva or vagina, vulvar and vaginal warmth such as burning, smearing, decreased lubrication during sexual activity and dyspareunia and postcoital bleeding, sexual reproduction such as decreased arousal and orgasm, and urinary problems such as incontinence, dysuria, frequent stopping and urgency. It contains sections (3). Approximately 50% of postmenopausal women are greatly affected in terms of both quality of life and vital functionality (4,5). Topical hormonal therapy is normally considered standard treatment for postmenopausal women. It ensures the epithelial integrity of women and the restoration and vaginal proliferation of the vaginal flora. Prescription of topical risks should also be avoided in patients with breast cancer, susceptible tumors and a history of thromboembolism; This situation emphasizes the necessity of treatment alternatives (6,7). Lubricants and moisturizers are options to help with drying, but sufficient data to screen for effectiveness have not been published (7). It is another alternative to ospemifene and breaks down the divisions depending on your hypoestrogen (8). Fractional CO 2 laser is an emerging treatment option for vaginal care, especially for women with contraindications to hormone therapy. Fractional CO 2 laser treatment consists of two or three sessions, and treatment responses only occur after a period of 20 weeks (9). Another treatment approach is pelvic floor exercises. Pelvic floor muscle training (PFMT) was first described as an effective method of urinary incontinence management by Arnold Kegel in 1948 (10). Although Kegel reports reported over 84% recovery rates for patients after PFMT, it remained the first-stage treatment approach until the 1980s. Following this payment, women's incontinence, health and sports opportunities, the cost of surgeries, the paths opened by the surgical route, services and the permanent deterioration of the recurrences that occur after surgery, and the interest in conservative treatments also come (11). In many systematic reviews, PFMT is considered to be the first step in the treatment of urinary incontinence (12,13). A recent single-arm feasibility study found a 12-week pelvic floor muscle training (PFMT) program, a normal symptom of postmenopausal bleeding with urinary incontinence and significant bursts. After the intervention, increased secretions in normal walls, thicker vaginal epithelial cells, and improvement in vaginal color were achieved. In other words, postmenopausal pelvic floor exercises increase vaginal secretions and restore normal size (14).

The purpose of this process is; To investigate the normal and sexual health status of pelvic floor exercises after menopause. In addition, generally normal behaviors were evaluated by observing them subjectively (9,15). In our study, we plan to evaluate normal dryness, which is one of the normal conditions, using the Schirmer Test. Additionally, our study will be the first to evaluate normal dryness of a lens.

ELIGIBILITY:
Inclusion Criteria:

* Having applied to Istanbul Training and Research Hospital, Gynecology and Obstetrics Polyclinic
* Being literate
* Volunteering to participate in the study
* Amenorrhea for 12 months
* Being sexually active
* BMI < 35
* Mini Mental Test Score threshold value for individuals over 65 years of age is 24

Exclusion Criteria:

* Active vaginal infection
* Having a history of active malignancy and receiving radiotherapy and/or chemotherapy accordingly
* Having received Hormone Replacement Therapy within the last year,
* Use of local estrogen
* Coitus in the last two days
* Pelvic organ prolapse stage 2 or higher
* Having had mesh surgery
* Presence of a disease/medication that causes vaginal dryness (e.g. Sjögren's syndrome, Lichen planus, Lichen Sclerosis / use of antidepressants or antihistamines).

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 20 (Estimated)
Dates: Start 2024-01-13 (Actual); Primary Completion 2024-07-13 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Schirmer's Test | 5 minutes
  This test was developed to diagnose dry eye (16). In this study, the test will be used to evaluate vaginal dryness. Test strips (ERC) not impregnated with blue dye, 5 mm wide and 35 mm long, are used for the test. The strip will be placed in the vagina, above the Carunculae Hymenalis, by holding it with sterile forceps or by holding the very end of the strip. After the test strip placement is standardized in this way, time will be kept with a stopwatch. The test strip will be left in the vagina for 5 minutes. When the time is completed, the test strip will be removed immediately and the distance the vaginal wetness has progressed will be measured according to the values on the strip.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 3 minutes
  Visual Analog Scale (VAS) is used to convert some values that cannot be measured digitally into digital form. The two ends of a 100 mm line are marked by defining the two ends of the parameter to be evaluated and by asking the patient where their parts fit on this line by drawing a line or by using punctuation or signs. The distance between the point placed and the lowest end of the line (0 = no symptoms) is measured as '0' when they do not feel any symptoms, and '10' when they have the most severe symptom that continues throughout their life, and the numerical value change is the symptom. is showing. The severity of vaginal dryness, burning and dyspareunia will be evaluated via VAS.
Female Sexual Function Index (FSFI) | 10 minutes
  Female Sexual Function Index, Rosen et al. It was developed in 2000 to evaluate female sexual functions. The Likert-type scale, consisting of 19 items, has 6 sub-dimensions: desire, arousal, lubrication, orgasm, satisfaction and pain. It has been reported that the FSFI is a valid and reliable tool in the evaluation of sexual function of Turkish women.
Postmenopausal Sexuality Questionnaire (PMSQ) | 10 minutes
  PMSQ was developed in 2020 by Maria Josef Lima and colleagues (17) to measure sexual activity after menopause. The original language of the scale has been deleted and an English version is also available. The survey contains 36 items assessing sexual activity. Questions are answered according to ordinal Likert scales (0-5). The total cost of the survey is shown as 215, and the total score due to the presence of intermittent questions is 100 maximum. 0 indicates the worst sexual function, 100 indicates the best sexual function (0-100). The scale has 9 subdomains: self-image, quality of sexual life, sexual intimacy, desire, importance of sexual life, arousal, orgasm, satisfaction and effects of menopause.
Vaginal Daily Impact of Aging Scale (VDIAS) | 10 minutes
  To evaluate the impact of vaginal symptoms on individuals' functionality and well-being, Alison Huang et al. The "Daily Effect of Vaginal Aging Scale (VYGE Scale)" developed by A.Ş. will be used. This scale comprehensively evaluates the impact of menopause-specific vaginal symptoms on daily living activity, emotional state, sexual health, and body image. The average score and total score can be calculated separately for the 4 subsections of the scale. While the scale subdomain scores vary between 0-4, the scale total score varies between 0-16. High scores obtained with the scale reflect the negative impact of vaginal symptoms on health-related quality of life.
Disturbing Pelvic Floor Inventory-20 | 10 minutes
  In order to measure the presence of pelvic floor symptoms and how much these symptoms bother the person, Toprak Celenay Ş. et al. "Pelvic Floor Distress Inventory-20" (PFDE-20), whose validity and reliability in Turkish has been demonstrated by , will be used. This scale is among the most commonly used tools to measure pelvic organ prolapse, urinary and colorecto-anal problems that may develop due to pelvic floor dysfunction, and the degree of discomfort associated with these symptoms. A total of 20 items belonging to 3 subdomains: "Pelvic Organ Prolapse Distress Inventory-, "Colorectal-Anal Distress Inventory-8" and "Urinary Distress Inventory-6" In the scale consisting of one item, the presence of pelvic floor symptoms is questioned and, if present, how much this symptom bothers the person is scored between 1-4, from "unimportant" to "very much".
Evaluation of Pelvic Floor Muscle Strength | 5 minutes
  Pelvic floor muscle strength is measured manually by asking the person to squeeze the index and middle fingers inserted into the vagina. This is a subjective method. The strength of the contraction felt around the finger is scored according to the Modified Oxford Scale created by Laycock and Chiarelli in 1989. In the digital palpation method, in addition to muscle strength, endurance, number of repetitions, speed and time are also measured using the 'PERFECT' system. The PERFECT system was created by Laycock and Jerwood in 2001, based on the Oxford scale (24).

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Gülşah KÜRNE, MsC, Study Chair — Hacettepe University
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No